CLINICAL TRIAL: NCT02966938
Title: Visual Recognition of Allergens by Allergic Patients and/or Their Parents
Acronym: REVIALL
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-048
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Nut Allergy; Peanut Allergy
MeSH Terms: conditions — Nut Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nut allergic patients: Allergic patient and their family with allergy to peanut or other tree nuts that are in elimination diet.

SUMMARY:
Food allergies are constantly increasing. Peanut and nut allergies are a major cause of allergic reactions. Diagnosed patients are also at risk, because 27% of the patients that had an allergic reaction have another one in the following year with the same food, despite a real improvement in industrial products labeling.

The investigators have observed in the allergy Unit that patients (and/or their family) following an elimination diet, sometimes since several years, use very strict elimination strategies. Those strategies sometimes lead to incapacities to recognize the allergens. Yet, a good identification of the allergen is the key to a successful elimination and the non-identification a known risk factor.

Ferdman shown in 2006 that 27% of the patients didn't recognize the allergen there were allergic to. However, this is a US study, and geographical specificities have an impact on food consumption and culture. Food allergology needs to take those two elements into account. For example, in France, a single food can have two names. It is the case of peanut, which can be called "arachide", or more frequently "cacahuète".

The goal of the study is to observe patient aptitudes to recognize peanut (and the association between the two names) and other nuts available in France and define by the European law, using a plate with various food samples in seed or in shell.

Thus, patients in care at the allergy Unit of Saint Vincent Hospital of Lille (France) and their families were surveyed with a standardized procedure at the beginning of their therapeutic education and their capacity to recognize various nuts, to identify peanut ("cacahuète" or "arachide") and to associate the two words "cacahuète" and "arachide" was assessed. It is a standard procedure in therapeutic education, and the responses have been systematically entered in the medical record.

The main objective of this study is to describe peanut or nut allergic patient capacity (adult, children and/or the family) to visually identify the foods there are allergic to.

The secondary objective of this study is to describe the capacity of patient that describe themselves as allergic to "arachide" to associate this word to the word "cacahuète".

ELIGIBILITY:
Inclusion Criteria:

* Peanut or nut allergy
* Following an elimination diet since at least 3 months
* Results obtained at the beginning of a therapeutic education started from 2013 to 2015

Exclusion Criteria:

* Patients opposed to enter the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their family with peanut or other nuts allergies followed in the allergy Unit of Saint Vincent Hospital of Lille (France) from 2013 to 2015, that are following an elimination diet and beginning a therapeutic education.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of patient that can visually identify the foods there are allergic to. | At inclusion

SECONDARY OUTCOMES:
number of patients presenting themselves as allergic to "arachide" knowing it is a synonym of "cacahuète" | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sauvage, MD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No